CLINICAL TRIAL: NCT06327568
Title: Anal Cancer and/or Precancer Screening: Performance Analysis of the BD Onclarity HPV Assay on Anal Specimens
Brief Title: Anal Cancer and/or Precancer Screening: Performance Analysis of the BD Onclarity™ HPV Assay on Anal Specimens
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1663
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Anal Intraepithelial Neoplasia 2; Anal Intraepithelial Neoplasia 1; Anal Cancer; High-Risk Cancer
Keywords: anal cancer; Human papillomavirus (HPV) infection; PCR genotyping; AIN 2
MeSH Terms: conditions — Anus Neoplasms; Papillomavirus Infections; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — anal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case patients: Histological-confirmed high-grade anal intraepithelial neoplasia (AIN2+ and 3+) and invasive cancer; patients with macroscopic anal lesion.
- Control patients: Histological-confirmed low-grade anal intraepithelial neoplasia (AIN1), and subjects at high-risk for anal cancers, including: Immunocompromised subjects (patients with HIV infection, or taking immunosuppressive drugs, or post-organ transplantation); Men who have sex with men (MSM); Women aged at least 40 years with a history of CIN2+ and/or vulvar cancer; Subjects affected by anal and/or peri-anal localizations of Crohn's disease.

SUMMARY:
Human papillomavirus (HPV) infection has been implicated as a necessary cause for the development of the majority of anogenital neoplasms which represent approximately 95% of anal tumors. Persistent high risk HR-HPV infection promotes progression from intraepithelial lesions high-grade squamous anal tumors (AIN) (H-SIL) to invasive anal tumors.

The diagnosis of AIN is made by cytology or biopsy during routine examinations. To date, no HPV test has been clinically validated for anal specimens and none are available in the molecular diagnostics market for this purpose.

The performance analysis of an HPV Test with simultaneous genotyping on anal samples could implement anal cancer screening without an invasive procedure and with one simple approach.

DETAILED DESCRIPTION:
Anal cancer is a rare disease in the general population, but its incidence is higher in certain at-risk groups, such as immunosuppressed individuals, including those with HIV infections and post-organ transplantation patients, men who have sex with men, and women with HPV-related lower genital tract dysplasia or cancer.

A squamous intraepithelial anal lesion is the dysplastic growth of squamous epithelial cells in the transition zone of the anal canal. This lesion is pre-malignant and can progress to anal squamous cell carcinoma if left untreated.

Human papillomavirus (HPV) infection has been implicated as the necessary cause for the development of the majority of anogenital malignancies accounting for approximately 95% of anal cancers. Persistent infection with HR-HPV promotes progression from high-grade squamous intraepithelial lesions (H-SIL) to invasive anal cancers. In the anal canal, low-grade intraepithelial lesion LSIL correlates with anal intraepithelial neoplasia (AIN)-1 or anal condyloma, while high grade squamous intraepithelial lesion HSIL correlates with AIN-2 and AIN-3.

Prevalence of H-SIL is around 40 to 50%. Progression from H-SIL to anal cancer is about 1/250 per year in HIV-positive MSM and 1/5000 per year in HIV-negative MSM, respectively.

The diagnosis of AIN is made from cytology or biopsy during routine examinations.

Up to date, different guidelines for anal cancer screening have been proposed but are not uniform. These include 1) digital ano-rectal examination, useful in unrecognized but symptomatic subjects, and 2) anal cytology, useful in asymptomatic subjects, only if high-resolution anoscopy is available.

These observations support the need to implement screening to prevent anal precancers and cancers.

At this moment, no HPV assay has been validated for anal specimens, and none is available in the molecular diagnostics market.

Validation of HPV typing methods on anal specimens could implement anal cancer screening without an invasive procedure and with an easy approach for the patient.

The BD Onclarity™ HPV Assay (BD Diagnostics, Sparks, USA) is a real-time polymerase chain reaction PCR assay that detects type-specific genomic DNA. The target of the assay is the E6 and E7 HPV genes. It simultaneously detects all 14 high-risk HPV types and can provide an "extended" genotype information on six individual genotypes (HPV 16, 18, 31, 45, 51 and 52), and in three distinct groups (33 and 58; 56, 59 and 66; and 35,39 and 68). Briefly, the DNA was extracted using BD FOX™ magnetic particles and the eluate-containing DNA was used to set up three PCR genotyping reactions: G1 detects HPV 16, HPV 18 and HPV 45 plus the internal beta globin control; G2 detects HPV 31, HPV 33_58 and HPV 56_59_66 plus the internal beta globin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years old
* Subjects with histological-confirmed high-grade anal intraepithelial neoplasia (AIN2+) or anal invasive cancer
* Subjects with histological-confirmed low-grade anal intraepithelial neoplasia (AIN1)
* Subjects at high-risk for anal cancers, including:

  1. Immunocompromised subjects (patients with HIV infection, or taking immunosuppressive drugs, or post-organ transplantation)
  2. Men who have sex with men (MSM)
  3. Women aged at least 40 years with a history of cervical intraepithelial neoplasia CIN2+ and/or vulvar cancer
  4. Subjects affected by anal and/or peri-anal localizations of Crohn's disease
* Subjects undergoing colorectal cancer screening
* Signed written consent.

Exclusion Criteria:

* Refuse to sign written consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who come at the European Institute of Oncology at high risk of anal cancer undergoing cancer screening anal, colorectal, or on an outpatient basis for HPV-related pathologies.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2029-06-17 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of BD Onclarity HPV assay for HPV detection and genotyping in case/control patients. | 4 years
  To evaluate to use of BD Onclarity HPV assay for HPV detection and genotyping from the anus, without endoscope. This study aims to enroll 100 cases and 100 controls to evaluate the performance of the Onclarity test in detecting the presence of HPV in anal swab samples that will be placed in a Thin Prep vial (Hologic), in order to perform cytology and the BD Onclarity assay, a qualitative target-amplification test based on RT-PCR and fluorescent probe technology to detect E6 and E7 DNA regions of the HPV genome; Onclarity provides genotyping information on six individual genotypes (HPV 16, 18, 31, 45, 51 and 52) and reports the remaining HPV genotypes in three distinct groups (33/58, 35/39/68, and 56/59/66). The assay has an internal human beta-globin (HBB) gene control for sample adequacy and assay performance. Sensitivity, specificity of the Onclarity test will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of Oncology, Milan, Italy